CLINICAL TRIAL: NCT04518163
Title: Bakri Balloon Tamponade Plus Intravenous Tranexamic Acid During Cesarean Delivery for Placenta Previa: a Randomized Double-blind Controlled Trial
Brief Title: Bakri Balloon Plus Tranexamic Acid During Cesarean Delivery for Placenta Previa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/279/7/19
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Bakri balloon was inserted into the lower uterine segment through the uterine incision by passing the balloon shaft through the cervix with an assistant pulling vaginally plus 1gm tranexamic acid by intravenous infusion
  Interventions: Drug: Tranexamic Acid; Device: Bakri Balloon
- control group (Active Comparator): Bakri balloon was inserted into the lower uterine segment through the uterine incision by passing the balloon shaft through the cervix with an assistant pulling vaginally plus saline by intravenous infusion
  Interventions: Drug: placebo to TA; Device: Bakri Balloon

INTERVENTIONS:
Drug: Tranexamic Acid — Intravenous 1 gm tranexamic acid in 100 ml saline by slow infusion before skin incision
  Other Names: TA
  Arms: study group
Drug: placebo to TA — Intravenous 110 ml saline by slow infusion before skin incision
  Other Names: saline
  Arms: control group
Device: Bakri Balloon — Bakri balloon was inserted into the lower uterine segment through the uterine incision by passing the balloon shaft through the cervix with an assistant pulling vaginally
  Other Names: BBT

SUMMARY:
Objective to investigate the effect of adjunctive intravenous tranexamic acid (TA) on blood loss during cesarean section (CS) in patients with placenta previa undergone Bakri balloon tamponade

DETAILED DESCRIPTION:
Placenta previa (PP) is an obstetric condition that is closely linked with massive obstetric hemorrhage with a varied incidence about once in every 200 live births. It is considered one of the causes of the increased need for blood transfusion and cesarean hysterectomy. PPH due to PP typically starts during cesarean section (CS) in the placental bed, at the lower uterine segment mostly after placental separation. Proceeding for cesarean hysterectomy can be the only effective line of management in spite of the associated high morbidity rate.

Tranexamic acid is a lysine analog which acts as an antifibrinolytic via competitive inhibition of the binding of plasmin and plasminogen to fibrin. The rationale for its use in the reduction of blood loss depending on the implication of the coagulation and fibrinolysis processes implicated in the control of PPH. However, concerns about possible thromboembolic events with parenteral administration of TA have stimulated increasing interest in its topical use.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing elective cesarean delivery for complete placenta previa which not respond uterotonic and simple hemostatic maneuvers like placental bed hemostatic sutures

Exclusion Criteria:

* patients with the high possibility of morbid adherent placenta
* those presented with severe antepartum hemorrhage
* Patients with cardiac, hepatic, renal, or thromboembolic disease;
* hypersensitivity or contraindications of use of tranexamic acid
* patient refuses to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women undergoing elective cesarean delivery for complete placenta previa
Enrollment: 140 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
mean Blood loss after placental separation | 30 minutes
  by using weight of soaked towels (weight of soaked towel - weight of dry towel) and amount of blood in suction set

SECONDARY OUTCOMES:
Number of Participants with postpartum hemorrhage | 12 hours
  number pf participants with blood loss > 1000ml
The number of participant needed of extra surgical maneuvers | 30minutes
  Calculation of the number of participant needed of extra surgical maneuvers like internal iliac artery ligation

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No